CLINICAL TRIAL: NCT03049514
Title: Study of Arterial Recanalization of the Central Retinal Artery Occlusions
Acronym: RECANAL
Status: Completed | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: MOA_2016_22
Record Dates: First submitted 2017-02-08; First posted 2017-02-10 (Actual); Last update posted 2022-04-14 (Actual); Status verified 2022-04

CONDITIONS: Central Retinal Artery Occlusion
Keywords: Thrombolysis; Recanalization; Dynamic retinal angiography
MeSH Terms: conditions — Retinal Artery Occlusion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Central retinal artery occlusions (CRAO) are the equivalent of an ischemic stroke (IS) at the retinal level. They share the same risk factors and common pathology. Their incidence is lower (8.5 / 100,000) and the functional prognosis is unfavorable in 80% of cases with visual acuity (VA) <1/10. The diagnosis of an CRAO is clinically based on the sudden occurrence of a decrease in deep visual acuity with fundamentally signs of reactive ischemia. There is no data on early retinal arterial recanalization after CRAO, nor on the relationship between early recanalization (spontaneous or post-thrombolysis) and visual prognosis.

ELIGIBILITY:
Inclusion Criteria:

* Central Retinal Artery Occlusion ≤ 24 hours

Exclusion Criteria:

* Retinal Dynamic angiography not performed within 48 hours of onset of symptoms
* Occlusion of a branch of the central retinal artery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients referred for an central retinal artery occlusion
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2016-12-23 (Actual); Primary Completion 2022-04-02 (Actual); Study Completion 2022-04-02 (Actual)

PRIMARY OUTCOMES:
Dynamic retinal angiography data at 24 hours (+/- 24 hours) | 24 hours (+/- 24 hours) following the beginning of symptoms
  Proportion of patients with early arterial recanalization.The recanalization rate will be compared between thrombolysed patients and non-thrombolysed patients

CONTACTS AND LOCATIONS:
Overall Officials: Michaël Obadia, MD, Principal Investigator — Fondation A de Rothschild
Locations (1):
- Fondation ophtalmique Adolphe de Rothschild, Paris, France

REFERENCES:
- [Derived] Abdelmassih Y, Mauget-Faysse M, Seners P, Milea D, Hallali G, Guillaume J, Lecler A, Vignal C, Le Mer Y, Paques M, Bonnin S, Obadia M. Early reperfusion in patients with acute retinal artery occlusion: A multicenter prospective study. Int J Stroke. 2025 Mar;20(3):338-346. doi: 10.1177/17474930241306692. Epub 2024 Dec 24. PMID 39614619